CLINICAL TRIAL: NCT05963087
Title: Cetuximab in Combination With Dabrafenib and Tislelizumab in BRAF Mutated Treatment of Advanced Colorectal Cancer: a Prospective, Exploratory, Phase II Clinical Study
Brief Title: Cetuximab in Combination With Dabrafenib and Tislelizumab in BRAF Mutated Treatment of Advanced Colorectal Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Wangxia LV, MD, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Braf-001
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Advanced Colorectal Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced CRC (Experimental): Patients with BRAF Mutated Advanced CRC were given Cetuximab in Combination With Dabrafenib and Tislelizumab
  Interventions: Drug: Cetuximab Dabrafenib Tislelizumab

INTERVENTIONS:
Drug: Cetuximab Dabrafenib Tislelizumab — Dabrafenib 150mg，BID, Cetuximab 250mg/m2, Tislelizumab 200mg Treatment every three weeks

SUMMARY:
To explore the efficacy and safety of Cetuximab in combination with dabrafenib and Tislelizumab in BRAF mutated treatment of advanced colorectal cancer

DETAILED DESCRIPTION:
Due to Encorafenib has not been marketed in China, it is difficult to benefit patients, and there are no reported studies of Dabrafenib, also a BRAF inhibitor, in combination with anti-EGFR monoclonal antibody and immunotherapy in BRAF mutated mCRC. Therefore, we intend to use Dabrafenib in combination with cetuximab and Tislelizumab in the treatment of BRAF V600E mutated patients with advanced colorectal cancer to observe the initial efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histopathological diagnosis of advanced colorectal cancer; 2. Previous first-line standard treatment failed or could not tolerate first-line standard treatment; 3. BRAF V600E mutation (NGS or ARMS-PCR assay); 4.18 years old≤ Age≤75 years old; 5. PS score 0-1; 6. At least one measurable or evaluable lesion according to RECIST v1.1; 7. Baseline color Doppler ultrasound: left ventricular ejection fraction (LVEF) ≥60%; 8. Has adequate organ and bone marrow function; 9. Expected survival ≥12 weeks 10. Female subjects of childbearing age or male subjects whose sexual partner is a female of childbearing age are required to take effective contraceptive measures throughout the treatment period and for 6 months after the treatment period 11. Sign a written informed consent and be able to comply with the visit and related procedures required by the program;

Exclusion Criteria:

* 1. Malignant diseases other than colorectal cancer diagnosed within 5 years prior to first administration (excluding radical treatment)Carcinomas in situ with sexual resection); 2. Currently participating in the intervention clinical study treatment, or receiving other study drugs or using study devices within 4 weeks before the first dose; 3. Previous treatment with BRAF inhibitors, MEK inhibitors, anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs, or drugs that target another stimulus or synergically inhibit T cell receptors (e.g., CTLA-4, OX-40, CD137); 4. Received systemic systemic treatment with Chinese patent drugs with anti-tumor indications or immunomodulatory drugs (including thymosin, interferon, interleukin, except for local use to control pleural fluid) within 2 weeks before the first administration; 5. An active autoimmune disease requiring systemic treatment (e.g. with disease-modifying drugs, glucocorticoids, or immunosuppressants) has occurred within 2 years prior to initial administration. Replacement therapies (such as thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy; 6. Were receiving systemic glucocorticoid therapy (excluding topical glucocorticoids by nasal spray, inhalation, or other route) or any other form of immunosuppressive therapy within 7 days prior to initial administration of the study 7. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation 8. Known allergy to any monoclonal antibody formulation ingredient (grade 3 or above allergic reaction) 9. Has not fully recovered from toxicity and/or complications caused by any intervention before starting treatment (i.e., ≤ grade 1 or baseline, excluding weakness or hair loss); 10. Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive); 11. Untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected greater than the upper limit of normal value in the laboratory of the study center); 12. Active HCV-infected subjects (HCV antibody positive and HCV-RNA levels above the lower limit of detection); 13. Received live vaccine within 30 days prior to the first dose (cycle 1, day 1); 14. Pregnant or lactating women; 15. The presence of any serious or uncontrolled systemic disease 16. Medical history or evidence of disease that may interfere with test results, prevent participants from fully participating in the study, abnormal treatment or laboratory test values, or other conditions that the investigator considers unsuitable for enrollment The Investigator considers other potential risks unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 12 months
  CR + PR rate according to the RECIST version 1.1 guidelines.

SECONDARY OUTCOMES:
Progression Free Survival (PFS） | up to 12 months
  To assess the efficacy of Surufatinib Combine With Immunotherapy and Chemotherapy as second-line therapy to Advanced CRC, patients by assessment of progression free survival (PFS) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
Overall survival time | up to 36 months
  OS was calculated from the date of pharmacy to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Wangxia Lv, Principal Investigator — Zhejiang Cancer Institute & Hospital
Locations (1):
- Zhejiang Cancer Institute & Hospital, Hangzhou, Zhejing, China